CLINICAL TRIAL: NCT01301625
Title: A Prospective Single Arm Clinical Trial Evaluating the MitraClip System in Australia and New Zealand
Brief Title: MitraClip System in Australia and New Zealand
Acronym: MitraClipANZ
Status: Terminated | Type: Observational
Why Stopped: As recruitment rate was lower than anticipated
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: Protocol #M10-001
Record Dates: First submitted 2011-02-04; First posted 2011-02-23 (Estimated); Results first posted 2018-10-22 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Mitral Regurgitation
Keywords: MitraClip; mitral regurgitation (MR); mitral valve insufficiency; percutaneous mitral valve repair; congestive heart failure
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- MitraClip Implant: Eligible patients undergoing a MitraClip procedure in Australia and New Zealand
  Interventions: Device: MitraClip Implant

INTERVENTIONS:
Device: MitraClip Implant — Percutaneous mitral valve repair using MitraClip implant.
  Other Names: MitraClip System; MitraClip Delivery System; Steerable Guide Catheter

SUMMARY:
The primary objective of the MitraClip System Australia and New Zealand (ANZ) Clinical Trial is to gather real-world clinical and health-economic outcome data to support the long-term safety, efficacy and economic value of the MitraClip System in the continuum of therapies for treating MR. Specifically, the following clinical and economic data will be collected: New York Heart Association (NYHA) Functional Class, Six-Minute Walk Test (6MWT) distance, quality of life (QOL) information, echocardiographic measures of left ventricular size and function, and data associated with the index hospitalization, rehospitalizations, concomitant medications and discharge facility to support the MitraClip System economic analysis.

DETAILED DESCRIPTION:
The MitraClip System ANZ Clinical Trial is a prospective, observational, single arm, multicenter trial to evaluate the MitraClip device for the treatment of mitral regurgitation (MR). Patients will be enrolled at up to 15 investigational sites throughout Australia and New Zealand. Up to 150 patients will be enrolled. Patients will be considered enrolled when local or general anesthesia is administered for the MitraClip procedure. Patients will be followed at discharge, 30 days, 6 months, 12 months and 24 months.

Investigational sites will recruit consecutive patients who meet trial enrollment criteria. Until enrollment in the MitraClip System ANZ Clinical Trial is closed, all patients who undergo a procedure for placement of a MitraClip device at an investigational site should be enrolled in the MitraClip System ANZ Clinical Trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* MR ≥ 3+ .
* Transseptal catheterization and femoral vein access feasible.
* Placement of the MitraClip device on mitral leaflets feasible.
* Mitral valve orifice area ≥ 4.0 cm2.
* Written informed consent obtained.
* The patient agrees to return for follow-up visits.

Exclusion Criteria:

* Need for emergency surgery, other cardiac surgery.
* Coronary artery disease (CAD), atrial fibrillation (AF), other valve disease.
* Prior mitral valve repair surgery, mechanical prosthetic valve, or ventricular assist device (VAD).
* Active endocarditis or rheumatic heart disease; leaflets degenerated from endocarditis or rheumatic disease.
* Transesophageal echocardiography (TEE) contraindicated.
* Known hypersensitivity or contraindication to trial or procedure medications which cannot be managed medically.
* Currently participating in investigational drug trial or another device trial that has not yet completed the primary endpoint or that interferes with the MitraClip System ANZ Clinical Trial.
* Pregnant or planning pregnancy within next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients eligible to receive the MitraClip implant at the designated investigational sites in Australia and New Zealand.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2011-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Muller, MD, Principal Investigator — St Vincent's Hospital - Sydney, Australia; Jurgen Passage, FRACs, Principal Investigator — Sir Charles Gairdner Hospital, Perth, Australia
Locations (6):
- Australia (6):
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Macquarie University Hosptial, North Ryde, New South Wales
  - North Shore Private Hospital, St Leonards, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia

REFERENCES:
- [Background] Mauri L, Garg P, Massaro JM, Foster E, Glower D, Mehoudar P, Powell F, Komtebedde J, McDermott E, Feldman T. The EVEREST II Trial: design and rationale for a randomized study of the evalve mitraclip system compared with mitral valve surgery for mitral regurgitation. Am Heart J. 2010 Jul;160(1):23-9. doi: 10.1016/j.ahj.2010.04.009. PMID 20598968
- [Background] Whitlow PL, Feldman T, Pedersen WR, Lim DS, Kipperman R, Smalling R, Bajwa T, Herrmann HC, Lasala J, Maddux JT, Tuzcu M, Kapadia S, Trento A, Siegel RJ, Foster E, Glower D, Mauri L, Kar S; EVEREST II Investigators. Acute and 12-month results with catheter-based mitral valve leaflet repair: the EVEREST II (Endovascular Valve Edge-to-Edge Repair) High Risk Study. J Am Coll Cardiol. 2012 Jan 10;59(2):130-9. doi: 10.1016/j.jacc.2011.08.067. PMID 22222076
- [Background] Tamburino C, Ussia GP, Maisano F, Capodanno D, La Canna G, Scandura S, Colombo A, Giacomini A, Michev I, Mangiafico S, Cammalleri V, Barbanti M, Alfieri O. Percutaneous mitral valve repair with the MitraClip system: acute results from a real world setting. Eur Heart J. 2010 Jun;31(11):1382-9. doi: 10.1093/eurheartj/ehq051. Epub 2010 Mar 18. PMID 20299349
- [Background] Ussia GP, Barbanti M, Tamburino C. Feasibility of percutaneous transcatheter mitral valve repair with the MitraClip system using conscious sedation. Catheter Cardiovasc Interv. 2010 Jun 1;75(7):1137-40. doi: 10.1002/ccd.22415. PMID 20336809
- [Background] Jonsson A, Settergren M. MitraClip catheter-based mitral valve repair system. Expert Rev Med Devices. 2010 Jul;7(4):439-47. doi: 10.1586/erd.10.23. PMID 20583881
- [Background] Argenziano M, Skipper E, Heimansohn D, Letsou GV, Woo YJ, Kron I, Alexander J, Cleveland J, Kong B, Davidson M, Vassiliades T, Krieger K, Sako E, Tibi P, Galloway A, Foster E, Feldman T, Glower D; EVEREST Investigators. Surgical revision after percutaneous mitral repair with the MitraClip device. Ann Thorac Surg. 2010 Jan;89(1):72-80; discussion p 80. doi: 10.1016/j.athoracsur.2009.08.063. PMID 20103209
- [Background] Geidel S, Ostermeyer J, Lass M, Schmoeckel M. Complex surgical valve repair after failed percutaneous mitral intervention using the MitraClip device. Ann Thorac Surg. 2010 Jul;90(1):277-9. doi: 10.1016/j.athoracsur.2009.12.048. PMID 20609795
- [Background] Kalarus Z, Kukulski T, Lekston A, Streb W, Sikora J, Nadziakiewicz P, Gasior M, Polonski L, Zembala M. [Methodology and safety of transvascular reduction of severe ischaemic mitral insufficiency with MitraClip in high-surgical-risk patients - first three cases in Poland]. Kardiol Pol. 2010 Jun;68(6):729-35. Polish. PMID 20806217
- [Background] Lim DS, Kunjummen BJ, Smalling R. Mitral valve repair with the MitraClip device after prior surgical mitral annuloplasty. Catheter Cardiovasc Interv. 2010 Sep 1;76(3):455-9. doi: 10.1002/ccd.22547. PMID 20839359
- [Background] Ciobanu A, Bennett S, Azam M, Clark A, Vinereanu D. Incremental value of three-dimensional transoesophageal echocardiography for guiding double percutaneous MitraClip (R) implantation in a 'no option' patient. Eur J Echocardiogr. 2011 Feb;12(2):E11. doi: 10.1093/ejechocard/jeq118. Epub 2010 Sep 27. PMID 20876188
- [Background] Tamburino C, Imme S, Barbanti M, Mule M, Pistritto AM, Aruta P, Cammalleri V, Scarabelli M, Mangiafico S, Scandura S, Ussia GP. Reduction of mitral valve regurgitation with Mitraclip(R) percutaneous system. Minerva Cardioangiol. 2010 Oct;58(5):589-98. PMID 20948505
- [Background] Borgia F, Di Mario C, Franzen O. Adenosine-induced asystole to facilitate MitraClip placement in a patient with adverse mitral valve morphology. Heart. 2011 May;97(10):864. doi: 10.1136/hrt.2010.208132. Epub 2010 Oct 29. No abstract available. PMID 21036802
- [Background] Luk A, Butany J, Ahn E, Fann JI, St Goar F, Thornton T, McDermott L, Madayag C, Komtebedde J. Mitral repair with the Evalve MitraClip device: histopathologic findings in the porcine model. Cardiovasc Pathol. 2009 Sep-Oct;18(5):279-85. doi: 10.1016/j.carpath.2008.07.001. Epub 2008 Aug 13. PMID 18703359
- [Background] Herrmann HC, Kar S, Siegel R, Fail P, Loghin C, Lim S, Hahn R, Rogers JH, Bommer WJ, Wang A, Berke A, Lerakis S, Kramer P, Wong SC, Foster E, Glower D, Feldman T; EVEREST Investigators. Effect of percutaneous mitral repair with the MitraClip device on mitral valve area and gradient. EuroIntervention. 2009 Jan;4(4):437-42. doi: 10.4244/eijv4i4a76. PMID 19284064
- [Background] Feldman T, Kar S, Rinaldi M, Fail P, Hermiller J, Smalling R, Whitlow PL, Gray W, Low R, Herrmann HC, Lim S, Foster E, Glower D; EVEREST Investigators. Percutaneous mitral repair with the MitraClip system: safety and midterm durability in the initial EVEREST (Endovascular Valve Edge-to-Edge REpair Study) cohort. J Am Coll Cardiol. 2009 Aug 18;54(8):686-94. doi: 10.1016/j.jacc.2009.03.077. PMID 19679246
- [Background] Rogers JH, Yeo KK, Carroll JD, Cleveland J, Reece TB, Gillinov AM, Rodriguez L, Whitlow P, Woo YJ, Herrmann HC, Young JN. Late surgical mitral valve repair after percutaneous repair with the MitraClip system. J Card Surg. 2009 Nov-Dec;24(6):677-81. doi: 10.1111/j.1540-8191.2009.00901.x. Epub 2009 Jul 24. PMID 19682161
- [Background] Silvestry FE, Rodriguez LL, Herrmann HC, Rohatgi S, Weiss SJ, Stewart WJ, Homma S, Goyal N, Pulerwitz T, Zunamon A, Hamilton A, Merlino J, Martin R, Krabill K, Block PC, Whitlow P, Tuzcu EM, Kapadia S, Gray WA, Reisman M, Wasserman H, Schwartz A, Foster E, Feldman T, Wiegers SE. Echocardiographic guidance and assessment of percutaneous repair for mitral regurgitation with the Evalve MitraClip: lessons learned from EVEREST I. J Am Soc Echocardiogr. 2007 Oct;20(10):1131-40. doi: 10.1016/j.echo.2007.02.003. Epub 2007 Jun 13. PMID 17570634
- [Background] Herrmann HC, Rohatgi S, Wasserman HS, Block P, Gray W, Hamilton A, Zunamon A, Homma S, Di Tullio MR, Kraybill K, Merlino J, Martin R, Rodriguez L, Stewart WJ, Whitlow P, Wiegers SE, Silvestry FE, Foster E, Feldman T. Mitral valve hemodynamic effects of percutaneous edge-to-edge repair with the MitraClip device for mitral regurgitation. Catheter Cardiovasc Interv. 2006 Dec;68(6):821-8. doi: 10.1002/ccd.20917. PMID 17080467
- [Background] Feldman T, Foster E, Glower DD, Kar S, Rinaldi MJ, Fail PS, Smalling RW, Siegel R, Rose GA, Engeron E, Loghin C, Trento A, Skipper ER, Fudge T, Letsou GV, Massaro JM, Mauri L; EVEREST II Investigators. Percutaneous repair or surgery for mitral regurgitation. N Engl J Med. 2011 Apr 14;364(15):1395-406. doi: 10.1056/NEJMoa1009355. Epub 2011 Apr 4. PMID 21463154
- [Background] Ladich E, Michaels MB, Jones RM, McDermott E, Coleman L, Komtebedde J, Glower D, Argenziano M, Feldman T, Nakano M, Virmani R; Endovascular Valve Edge-to-Edge Repair Study (EVEREST) Investigators. Pathological healing response of explanted MitraClip devices. Circulation. 2011 Apr 5;123(13):1418-27. doi: 10.1161/CIRCULATIONAHA.110.978130. Epub 2011 Mar 21. PMID 21422390
- [Background] Siegel RJ, Biner S, Rafique AM, Rinaldi M, Lim S, Fail P, Hermiller J, Smalling R, Whitlow PL, Herrmann HC, Foster E, Feldman T, Glower D, Kar S; EVEREST Investigators. The acute hemodynamic effects of MitraClip therapy. J Am Coll Cardiol. 2011 Apr 19;57(16):1658-65. doi: 10.1016/j.jacc.2010.11.043. PMID 21492763
- [Background] Grayburn PA, Roberts BJ, Aston S, Anwar A, Hebeler RF Jr, Brown DL, Mack MJ. Mechanism and severity of mitral regurgitation by transesophageal echocardiography in patients referred for percutaneous valve repair. Am J Cardiol. 2011 Sep 15;108(6):882-7. doi: 10.1016/j.amjcard.2011.05.013. Epub 2011 Jul 7. PMID 21741608
- [Background] Nor Aripin KN, Sammons HM, Choonara I. Published pediatric randomized drug trials in developing countries, 1996-2002. Paediatr Drugs. 2010 Apr 1;12(2):99-103. doi: 10.2165/11316260-000000000-00000. PMID 20218746
- [Background] Auricchio A, Schillinger W, Meyer S, Maisano F, Hoffmann R, Ussia GP, Pedrazzini GB, van der Heyden J, Fratini S, Klersy C, Komtebedde J, Franzen O; PERMIT-CARE Investigators. Correction of mitral regurgitation in nonresponders to cardiac resynchronization therapy by MitraClip improves symptoms and promotes reverse remodeling. J Am Coll Cardiol. 2011 Nov 15;58(21):2183-9. doi: 10.1016/j.jacc.2011.06.061. PMID 22078424
- [Background] Conradi L, Treede H, Franzen O, Seiffert M, Baldus S, Schirmer J, Meinertz T, Reichenspurner H. Impact of MitraClip therapy on secondary mitral valve surgery in patients at high surgical risk. Eur J Cardiothorac Surg. 2011 Dec;40(6):1521-6. doi: 10.1016/j.ejcts.2011.03.007. Epub 2011 Apr 15. PMID 21497508
- [Background] Divchev D, Kische S, Paranskaya L, Schneider H, Rehders T, Ortak J, Akin I, Turan G, Turan CH, Steinhoff G, Noldge-Schomburg G, Nienaber CA, Ince H. In-hospital outcome of patients with severe mitral valve regurgitation classified as inoperable and treated with the MitraClip(R) device. J Interv Cardiol. 2012 Apr;25(2):180-9. doi: 10.1111/j.1540-8183.2011.00688.x. Epub 2011 Dec 21. PMID 22188385
- [Background] Franzen O, van der Heyden J, Baldus S, Schluter M, Schillinger W, Butter C, Hoffmann R, Corti R, Pedrazzini G, Swaans MJ, Neuss M, Rudolph V, Surder D, Grunenfelder J, Eulenburg C, Reichenspurner H, Meinertz T, Auricchio A. MitraClip(R) therapy in patients with end-stage systolic heart failure. Eur J Heart Fail. 2011 May;13(5):569-76. doi: 10.1093/eurjhf/hfr029. Epub 2011 Apr 6. PMID 21471146
- [Background] Gaemperli O, Moccetti M, Surder D, Biaggi P, Hurlimann D, Kretschmar O, Buehler I, Bettex D, Felix C, Luscher TF, Falk V, Grunenfelder J, Corti R. Acute haemodynamic changes after percutaneous mitral valve repair: relation to mid-term outcomes. Heart. 2012 Jan;98(2):126-32. doi: 10.1136/heartjnl-2011-300705. Epub 2011 Oct 7. PMID 21983251
- [Background] Pleger ST, Mereles D, Schulz-Schonhagen M, Krumsdorf U, Chorianopoulos E, Rottbauer W, Katus HA, Bekeredjian R. Acute safety and 30-day outcome after percutaneous edge-to-edge repair of mitral regurgitation in very high-risk patients. Am J Cardiol. 2011 Nov 15;108(10):1478-82. doi: 10.1016/j.amjcard.2011.06.069. Epub 2011 Sep 3. PMID 21890084
- [Background] Rudolph V, Knap M, Franzen O, Schluter M, de Vries T, Conradi L, Schirmer J, Treede H, Wegscheider K, Costard-Jackle A, Meinertz T, Reichenspurner H, Baldus S. Echocardiographic and clinical outcomes of MitraClip therapy in patients not amenable to surgery. J Am Coll Cardiol. 2011 Nov 15;58(21):2190-5. doi: 10.1016/j.jacc.2011.07.047. PMID 22078425
- [Background] Schillinger W, Athanasiou T, Weicken N, Berg L, Tichelbacker T, Puls M, Hunlich M, Wachter R, Helms HJ, Seipelt R, Schondube FA, Hasenfuss G. Impact of the learning curve on outcomes after percutaneous mitral valve repair with MitraClip and lessons learned after the first 75 consecutive patients. Eur J Heart Fail. 2011 Dec;13(12):1331-9. doi: 10.1093/eurjhf/hfr141. Epub 2011 Oct 24. PMID 22024027
- [Background] Treede H, Schirmer J, Rudolph V, Franzen O, Knap M, Schluter M, Conradi L, Seiffert M, Koschyk D, Meinertz T, Baldus S, Reichenspurner H. A heart team's perspective on interventional mitral valve repair: percutaneous clip implantation as an important adjunct to a surgical mitral valve program for treatment of high-risk patients. J Thorac Cardiovasc Surg. 2012 Jan;143(1):78-84. doi: 10.1016/j.jtcvs.2011.09.033. Epub 2011 Oct 27. PMID 22036261
- [Background] Ussia GP, Cammalleri V, Sarkar K, Scandura S, Imme S, Pistritto AM, Caggegi A, Chiaranda M, Mangiafico S, Barbanti M, Scarabelli M, Mule M, Aruta P, Tamburino C. Quality of life following percutaneous mitral valve repair with the MitraClip System. Int J Cardiol. 2012 Mar 8;155(2):194-200. doi: 10.1016/j.ijcard.2011.08.853. Epub 2011 Sep 28. PMID 21955607
- [Background] Chan PH, Di Mario C, Franzen O. Dissociation between anatomical and functional results after MitraClip implantation. Int J Cardiol. 2012 Mar 8;155(2):175-6. doi: 10.1016/j.ijcard.2011.10.047. Epub 2011 Nov 9. No abstract available. PMID 22078980
- [Background] Rogers JH, Bolling SF. Editorial comment: Surgery after MitraClip therapy: you can't win them all. Eur J Cardiothorac Surg. 2011 Dec;40(6):1526-8. doi: 10.1016/j.ejcts.2011.04.024. Epub 2011 Jun 12. No abstract available. PMID 21664143
- [Background] Turi ZG, Rosenbloom M. An option for the high-comorbidity patient with mitral regurgitation. J Am Coll Cardiol. 2012 Jan 10;59(2):140-2. doi: 10.1016/j.jacc.2011.09.049. No abstract available. PMID 22222077
- [Background] Altiok E, Becker M, Hamada S, Reith S, Marx N, Hoffmann R. Optimized guidance of percutaneous edge-to edge repair of the mitral valve using real-time 3-D transesophageal echocardiography. Clin Res Cardiol. 2011 Aug;100(8):675-81. doi: 10.1007/s00392-011-0296-1. Epub 2011 Mar 3. PMID 21369924
- [Background] Bergsland J, Mujanovic E, Elle OJ, Mirtaheri P, Fosse E. Minimally invasive repair of the mitral valve: technological and clinical developments. Minim Invasive Ther Allied Technol. 2011 Apr;20(2):72-7. doi: 10.3109/13645706.2011.554843. PMID 21417839
- [Background] Biner S, Perk G, Kar S, Rafique AM, Slater J, Shiota T, Hussaini A, Chou S, Kronzon I, Siegel RJ. Utility of combined two-dimensional and three-dimensional transesophageal imaging for catheter-based mitral valve clip repair of mitral regurgitation. J Am Soc Echocardiogr. 2011 Jun;24(6):611-7. doi: 10.1016/j.echo.2011.02.005. Epub 2011 Mar 23. PMID 21435839
- [Background] Buch MH, Trento A, Kar S. Is there a role for surgeons in transcatheter mitral valve procedures? Curr Opin Cardiol. 2011 Mar;26(2):99-105. doi: 10.1097/HCO.0b013e32834398a0. PMID 21297461
- [Background] Chiam PT, Ruiz CE. Percutaneous transcatheter mitral valve repair: a classification of the technology. JACC Cardiovasc Interv. 2011 Jan;4(1):1-13. doi: 10.1016/j.jcin.2010.09.023. PMID 21251623
- [Background] Cikirikcioglu M, Cherian S, Schussler O, Kalangos A. Regarding "The EVEREST II Trial: design and rationale for a randomized study of the Evalve MitraClip system compared with mitral valve surgery for mitral regurgitation". Am Heart J. 2011 Jul;162(1):e11-2; author reply e13. doi: 10.1016/j.ahj.2011.04.004. Epub 2011 Jun 12. No abstract available. PMID 21742074
- [Background] Cleland JG, Coletta AP, Freemantle N, Clark AL. Clinical trials update from the American College of Cardiology Meeting 2011: STICH, NorthStar, TARGET, and EVEREST II. Eur J Heart Fail. 2011 Jul;13(7):805-8. doi: 10.1093/eurjhf/hfr077. PMID 21712293
- [Background] Dixon SR, Grines CL, O'Neill WW. The year in interventional cardiology. J Am Coll Cardiol. 2010 May 18;55(20):2272-86. doi: 10.1016/j.jacc.2010.02.024. No abstract available. PMID 20466207
- [Background] Dudiy Y, Jelnin V, Ruiz CE. Percutaneous mitral valve treatment. Minerva Cardioangiol. 2011 Oct;59(5):507-18. PMID 21983311
- [Background] Farouque HM, Clark DJ. Percutaneous mitral valve leaflet repair for mitral regurgitation: NICE guidance. Heart. 2010 Mar;96(5):385-7. doi: 10.1136/hrt.2009.183269. No abstract available. PMID 20197362
- [Background] Feldman T, Cilingiroglu M. Percutaneous leaflet repair and annuloplasty for mitral regurgitation. J Am Coll Cardiol. 2011 Feb 1;57(5):529-37. doi: 10.1016/j.jacc.2010.10.012. PMID 21272742
- [Background] George JC, Varghese V, Dangas G, Feldman TE. Percutaneous mitral valve repair: lessons from the EVEREST II (Endovascular Valve Edge-to-Edge REpair Study) and beyond. JACC Cardiovasc Interv. 2011 Jul;4(7):825-7. doi: 10.1016/j.jcin.2011.05.010. No abstract available. PMID 21777895
- [Background] Goldberg SL, Feldman T. Percutaneous mitral valve interventions: overview of new approaches. Curr Cardiol Rep. 2010 Sep;12(5):404-12. doi: 10.1007/s11886-010-0130-9. PMID 20617412
- [Background] Hussaini A, Kar S. Percutaneous mitral valve repair: potential in heart failure management. Curr Heart Fail Rep. 2010 Mar;7(1):22-6. doi: 10.1007/s11897-010-0006-8. PMID 20425493
- [Background] Jilaihawi H, Hussaini A, Kar S. MitraClip: a novel percutaneous approach to mitral valve repair. J Zhejiang Univ Sci B. 2011 Aug;12(8):633-7. doi: 10.1631/jzus.B1101009. PMID 21796803
- [Background] Lam YY, Lee PW, Yong G, Yan BP. Investigational devices for mitral regurgitation: state of the art. Expert Rev Med Devices. 2011 Jan;8(1):105-14. doi: 10.1586/erd.10.52. PMID 21158545
- [Background] Maisano F, Godino C, Giacomini A, Denti P, Arendar I, Buzzatti N, Canna GL, Alfieri O, Colombo A. Clinical trial experience with the MitraClip catheter based mitral valve repair system. Int J Cardiovasc Imaging. 2011 Dec;27(8):1155-64. doi: 10.1007/s10554-011-9872-8. Epub 2011 Apr 19. PMID 21503702
- [Background] Maisano F, Alfieri O, La Canna G. Percutaneous mitral repair with the MitraClip. Ann Fr Anesth Reanim. 2011 May;30 Suppl 1:S33-7. doi: 10.1016/S0750-7658(11)70008-9. PMID 21703485
- [Background] Maisano F, Godino C, Giacomini A, Denti P, Buzzatti N, Arendar I, Colombo A, Alfieri O, La Canna G. Patient selection for MitraClip therapy impaired left ventricular systolic function. Minerva Cardioangiol. 2011 Oct;59(5):455-71. PMID 21983306
- [Background] Maisano F, La Canna G, Colombo A, Alfieri O. The evolution from surgery to percutaneous mitral valve interventions: the role of the edge-to-edge technique. J Am Coll Cardiol. 2011 Nov 15;58(21):2174-82. doi: 10.1016/j.jacc.2011.07.046. PMID 22078423
- [Background] Ong SH, Beucher H, Mueller R, Gerckens U, Boekstegers P. Percutaneous double-valve interventions for aortic stenosis and pure mitral regurgitation. Am J Cardiol. 2011 Sep 15;108(6):893-5. doi: 10.1016/j.amjcard.2011.05.017. Epub 2011 Jul 2. PMID 21726839
- [Background] Padala M, Keeling WB, Guyton RA, Thourani VH. Innovations in therapies for heart valve disease. Circ J. 2011;75(5):1028-41. doi: 10.1253/circj.cj-11-0289. Epub 2011 Apr 9. PMID 21478626
- [Background] Rogers JH, Franzen O. Percutaneous edge-to-edge MitraClip therapy in the management of mitral regurgitation. Eur Heart J. 2011 Oct;32(19):2350-7. doi: 10.1093/eurheartj/ehr101. Epub 2011 May 23. PMID 21606080
- [Background] Saroul C, Keller G, Benaissa M, Lehot JJ. [Anesthesia for minimally invasive cardiac procedure]. Ann Fr Anesth Reanim. 2011 May;30 Suppl 1:S38-43. doi: 10.1016/S0750-7658(11)70009-0. French. PMID 21703486
- [Background] Seeburger J, Katus HA, Pleger ST, Krumsdorf U, Mohr FW, Bekeredjian R. Percutaneous and surgical treatment of mitral valve regurgitation. Dtsch Arztebl Int. 2011 Dec;108(48):816-21. doi: 10.3238/arztebl.2011.0816. Epub 2011 Dec 2. PMID 22211148
- [Background] Taramasso M, Cioni M, Giacomini A, Michev I, Godino C, Montorfano M, Colombo A, Alfieri O, Maisano F. Emerging approaches of transcatheter valve repair/insertion. Cardiol Res Pract. 2010 Jul 25;2010:540749. doi: 10.4061/2010/540749. PMID 20811476
- [Background] Taylor J. The percutaneous approach to mitral valve repair. Eur Heart J. 2011 Feb;32(3):249-51. doi: 10.1093/eurheartj/ehq463. No abstract available. PMID 21285076
- [Background] Vahanian A, Himbert D, Brochet E, Messika-Zeitoun D. Percutaneous mitral valve repair: the beginning of the end or the end of the beginning? F1000 Med Rep. 2010 Mar 25;2:21. doi: 10.3410/M2-21. PMID 20948864
- [Background] Van Mieghem NM, Piazza N, Anderson RH, Tzikas A, Nieman K, De Laat LE, McGhie JS, Geleijnse ML, Feldman T, Serruys PW, de Jaegere PP. Anatomy of the mitral valvular complex and its implications for transcatheter interventions for mitral regurgitation. J Am Coll Cardiol. 2010 Aug 17;56(8):617-26. doi: 10.1016/j.jacc.2010.04.030. PMID 20705218
- [Background] Walenta K, Sinning JM, Werner C, Bohm M. Hotline update of clinical trials and registries presented at the at the European Society of Cardiology Congress in Paris 2011. Clin Res Cardiol. 2011 Nov;100(11):955-71. doi: 10.1007/s00392-011-0370-8. Epub 2011 Sep 30. PMID 21960419
- [Background] Yuksel UC, Kapadia SR, Tuzcu EM. Percutaneous mitral repair: patient selection, results, and future directions. Curr Cardiol Rep. 2011 Apr;13(2):100-6. doi: 10.1007/s11886-010-0158-x. PMID 21184204
- [Background] Altiok E, Paetsch I, Jahnke C, Brehmer K, Reith S, Becker M, Marx N, Hoffmann R. Percutaneous edge-to-edge mitral valve repair: assessment of immediate post-procedural treatment effect using color 3-dimensional transesophageal echocardiography and cardiac magnetic resonance imaging. J Am Coll Cardiol. 2011 Sep 6;58(11):e21. doi: 10.1016/j.jacc.2010.11.088. No abstract available. PMID 21884943
- [Background] Barbanti M, Ussia GP, Tamburino C. Percutaneous treatment of aortic stenosis and mitral regurgitation in the same patient: first human cases description. Catheter Cardiovasc Interv. 2011 Oct 1;78(4):650-5. doi: 10.1002/ccd.23015. Epub 2011 Jul 25. PMID 21793170
- [Background] Bekeredjian R, Mereles D, Pleger S, Krumsdorf U, Katus HA, Rottbauer W. Large atrial thrombus formation after MitraClip implantation: is anticoagulation mandatory? J Heart Valve Dis. 2011 Mar;20(2):146-8. PMID 21560812
- [Background] Conradi L, Treede H, Baldus S, Seiffert M, Blankenberg S, Reichenspurner H. [Treating mitral regurgitation: a surgical and interventional update]. Herz. 2011 Dec;36(8):677-85. doi: 10.1007/s00059-011-3531-7. German. PMID 21994032
- [Background] Franzen O, von Samson P, Dodge-Khatami A, Geffert G, Baldus S. Percutaneous edge-to-edge repair of tricuspid regurgitation in congenitally corrected transposition of the great arteries. Congenit Heart Dis. 2011 Jan-Feb;6(1):57-9. doi: 10.1111/j.1747-0803.2010.00428.x. PMID 21269414
- [Background] Franzen O, Seiffert M, Baldus S, Conradi L, Schirmer J, Kubik M, Meinertz T, Reichenspurner H, Treede H. Percutaneous mitral valve repair as a bail-out strategy for patients with severe mitral regurgitation after cardiac surgery. J Thorac Cardiovasc Surg. 2011 Jul;142(1):227-30. doi: 10.1016/j.jtcvs.2010.10.037. Epub 2011 Jan 17. No abstract available. PMID 21247591
- [Background] Ihlemann N, Franzen O, Jorgensen E, Hansen PB, Hassager C, Moller JE, Sondergaard L. Promising results after percutaneous mitral valve repair. Dan Med Bull. 2011 Jul;58(7):A4299. PMID 21722544
- [Background] Kische S, Nienaber C, Ince H. Use of four MitraClip devices in a patient with ischemic cardiomyopathy and mitral regurgitation: "zipping by clipping". Catheter Cardiovasc Interv. 2012 Nov 15;80(6):1007-13. doi: 10.1002/ccd.23431. Epub 2012 Jan 10. PMID 22120912
- [Background] Kluge JG, Hagendorff A, Pfeiffer D, Jurisch D, Tarr A. Active infective prosthetic endocarditis after percutaneous edge-to-edge mitral valve repair. Eur J Echocardiogr. 2011 Sep;12(9):710. doi: 10.1093/ejechocard/jer062. Epub 2011 Jul 23. No abstract available. PMID 21785123
- [Background] Madder RD, Safian RD, Gallagher M, Senter SR, Hanzel GS. The first report of transcatheter aortic valve implantation and percutaneous mitral valve repair in the same patient. JACC Cardiovasc Interv. 2011 Jul;4(7):824. doi: 10.1016/j.jcin.2011.05.009. No abstract available. PMID 21777894
- [Background] Mayr NP, Martin K, Hausleiter J, Brown A, Tassani P. Ventilation manoeuvres facilitate MitraClip placement. Heart. 2011 Oct;97(20):1717; author reply 1717. doi: 10.1136/heartjnl-2011-300587. Epub 2011 Jul 31. No abstract available. PMID 21807657
- [Background] Paranskaya L, Turan I, Kische S, Nienaber C, Ince H. Rapid pacing facilitates grasping and MitraClip implantation in severe mitral leaflet prolapse. Clin Res Cardiol. 2012 Jan;101(1):69-71. doi: 10.1007/s00392-011-0384-2. Epub 2011 Nov 19. No abstract available. PMID 22102101
- [Background] Surder D, Altwegg L, Hurlimann D, Felix C, Grunenfelder J, Corti R. Percutaneous double valve intervention. Eur Heart J. 2011 Mar;32(5):636. doi: 10.1093/eurheartj/ehq378. Epub 2010 Nov 23. No abstract available. PMID 21098555
- [Background] Van den Branden BJ, Post MC, Swaans MJ, Rensing BJ, Eefting FD, Plokker HW, Jaarsma W, Van der Heyden JA. Percutaneous mitral valve repair using the edge-to-edge technique in a high-risk population. Neth Heart J. 2010 Sep;18(9):437-43. doi: 10.1007/BF03091811. PMID 20862239
- [Background] Van den Branden BJ, Swaans MJ, Post MC, Rensing BJ, Eefting FD, Jaarsma W, Van der Heyden JA. Redo mitral valve clipping after partial clip detachment. JACC Cardiovasc Interv. 2010 Feb;3(2):251-2. doi: 10.1016/j.jcin.2009.09.018. No abstract available. PMID 20170885
- [Background] Zuern CS, Schreieck J, Weig HJ, Gawaz M, May AE. Percutaneous mitral valve repair using the MitraClip in acute cardiogenic shock. Clin Res Cardiol. 2011 Aug;100(8):719-21. doi: 10.1007/s00392-011-0324-1. Epub 2011 May 24. No abstract available. PMID 21607532
- [Background] Alfieri O, Denti P. Alfieri stitch and its impact on mitral clip. Eur J Cardiothorac Surg. 2011 Jun;39(6):807-8. doi: 10.1016/j.ejcts.2011.01.017. Epub 2011 Feb 25. No abstract available. PMID 21353584
- [Background] Asgar AW, Khairy P. Percutaneous repair or surgery for mitral regurgitation. N Engl J Med. 2011 Jul 7;365(1):90; author reply 91. doi: 10.1056/NEJMc1105564. No abstract available. PMID 21732844
- [Background] Gorman RC, Gillespie MJ, Gorman JH 3rd. Percutaneous repair or surgery for mitral regurgitation. N Engl J Med. 2011 Jul 7;365(1):90-1; author reply 91. doi: 10.1056/NEJMc1105564. No abstract available. PMID 21732843
- [Background] Murphy MO, Ahmed K, Athanasiou T. Surgery for chronic ischemic mitral regurgitation - which mitral intervention? Expert Rev Cardiovasc Ther. 2011 May;9(5):587-97. doi: 10.1586/erc.11.50. PMID 21615322
- [Background] Osorio J, Fuster V. Valve interventions-a word of caution. Nat Rev Cardiol. 2010 Jul;7(7):355. doi: 10.1038/nrcardio.2010.83. No abstract available. PMID 20577293
- [Background] Otto CM, Verrier ED. Mitral regurgitation--what is best for my patient? N Engl J Med. 2011 Apr 14;364(15):1462-3. doi: 10.1056/NEJMe1102013. Epub 2011 Apr 4. No abstract available. PMID 21463152
- [Background] Skipper ER, Accola KD, Sade RM. Must surgeons tell mitral valve repair candidates about a new percutaneous repair device that is only available elsewhere? Ann Thorac Surg. 2011 Oct;92(4):1163-9. doi: 10.1016/j.athoracsur.2011.04.096. No abstract available. PMID 21958761
- [Background] Thompson KA, Philip KJ, Simsir S, Schwarz ER. The new concept of ''interventional heart failure therapy'': part 2--inotropes, valvular disease, pumps, and transplantation. J Cardiovasc Pharmacol Ther. 2010 Sep;15(3):231-43. doi: 10.1177/1074248410369111. Epub 2010 Jul 1. PMID 20595625
- [Background] Vahanian A, Iung B. 'Edge to edge' percutaneous mitral valve repair in mitral regurgitation: it can be done but should it be done? Eur Heart J. 2010 Jun;31(11):1301-4. doi: 10.1093/eurheartj/ehq088. Epub 2010 Apr 11. No abstract available. PMID 20385570
- [Background] Vahanian A, Iung B, Himbert D, Nataf P. Changing demographics of valvular heart disease and impact on surgical and transcatheter valve therapies. Int J Cardiovasc Imaging. 2011 Dec;27(8):1115-22. doi: 10.1007/s10554-011-9804-7. Epub 2011 Feb 24. PMID 21347599
- [Background] van den Heuvel AF, Alfieri O, Mariani MA. MitraClip in end-stage heart failure: a realistic alternative to surgery? Eur J Heart Fail. 2011 May;13(5):472-4. doi: 10.1093/eurjhf/hfr038. No abstract available. PMID 21505057
- [Background] Altiok E, Becker M, Hamada S, Grabskaya E, Reith S, Marx N, Hoffmann R. Real-time 3D TEE allows optimized guidance of percutaneous edge-to-edge repair of the mitral valve. JACC Cardiovasc Imaging. 2010 Nov;3(11):1196-8. doi: 10.1016/j.jcmg.2010.07.010. No abstract available. PMID 21071008
- [Background] Avanzini A, Donzella G, Libretti L. Functional and structural effects of percutaneous edge-to-edge double-orifice repair under cardiac cycle in comparison with suture repair. Proc Inst Mech Eng H. 2011 Oct;225(10):959-71. doi: 10.1177/0954411911414803. PMID 22204118
- [Background] Delgado V, Kapadia S, Marsan NA, Schalij MJ, Tuzcu EM, Bax JJ. Multimodality imaging before, during, and after percutaneous mitral valve repair. Heart. 2011 Oct;97(20):1704-14. doi: 10.1136/hrt.2011.227785. No abstract available. PMID 21949284
- [Background] Ewe SH, Klautz RJ, Schalij MJ, Delgado V. Role of computed tomography imaging for transcatheter valvular repair/insertion. Int J Cardiovasc Imaging. 2011 Dec;27(8):1179-93. doi: 10.1007/s10554-011-9830-5. Epub 2011 Feb 26. PMID 21359516
- [Background] Lin BA, Forouhar AS, Pahlevan NM, Anastassiou CA, Grayburn PA, Thomas JD, Gharib M. Color Doppler jet area overestimates regurgitant volume when multiple jets are present. J Am Soc Echocardiogr. 2010 Sep;23(9):993-1000. doi: 10.1016/j.echo.2010.06.011. Epub 2010 Aug 8. PMID 20696550
- [Background] Pedrazzini GB, Klimusina J, Pasotti E, Moccetti T, Faletra FF. Complications of percutaneous edge-to-edge mitral valve repair: the role of real-time three-dimensional transesophageal echocardiography. J Am Soc Echocardiogr. 2011 Jun;24(6):706.e5-7. doi: 10.1016/j.echo.2010.08.017. Epub 2010 Sep 26. PMID 20870392
- [Background] Siegel RJ, Luo H, Biner S. Transcatheter valve repair/implantation. Int J Cardiovasc Imaging. 2011 Dec;27(8):1165-77. doi: 10.1007/s10554-011-9833-2. Epub 2011 Feb 23. PMID 21344247
- [Background] Franzen O, Baldus S, Rudolph V, Meyer S, Knap M, Koschyk D, Treede H, Barmeyer A, Schofer J, Costard-Jackle A, Schluter M, Reichenspurner H, Meinertz T. Acute outcomes of MitraClip therapy for mitral regurgitation in high-surgical-risk patients: emphasis on adverse valve morphology and severe left ventricular dysfunction. Eur Heart J. 2010 Jun;31(11):1373-81. doi: 10.1093/eurheartj/ehq050. Epub 2010 Mar 10. PMID 20219746
- [Background] Yong ZY, Bouma BJ, Koch KT, Baan J. Immediate reduction of mitral regurgitation by percutaneous mitral valve repair with the MitraClip(R). Neth Heart J. 2010 Dec;18(12):606. doi: 10.1007/s12471-010-0843-9. No abstract available. PMID 21301624

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventy eight (78) patients who met trial enrollment criteria were enrolled at 6 investigational sites throughout Australia and New Zealand. Enrollment period was November 24, 2011 to June 15, 2014.
Period: Overall Study
Arm/Group | MitraClip Implant
Started | 78
Completed | 43
Not Completed | 35
Not completed — Death | 5
Not completed — Not Due | 21
Not completed — Expected | 8
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 54
Region of Enrollment [Number; unit: participants] — Total patient population was enrolled from Australia. No patients were enrolled from New Zealand. The study recruitment rate was lower than anticipated.
  participants
    Australia | 78

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Death (Kaplan-Meier Analysis)
Description: Clinical Endpoint.
  * Cardiac death is defined as any death in which a cardiac cause cannot be excluded. (This includes but is not limited to acute myocardial infarction, cardiac perforation/pericardial tamponade, arrhythmia or conduction abnormality,cerebrovascular accident within 30 days of the procedure or cerebrovascular accident suspected of being related to the procedure, death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery.)
  * Non-cardiac death is defined as a death not due to cardiac causes (as defined above).
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 78
percentage of participants | 0.0

2. Primary Outcome: Percentage of Participants Experiencing Death (Kaplan-Meier Analysis)
Description: as for outcome 1
Time Frame: 30 days
Population: Two patient were lost to follow-up at the 30-day time point and were not included in the "at risk" population in the Kaplan-Meier freedom from mortality analysis.
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 76
percentage of participants | 0.0

3. Primary Outcome: Percentage of Participants Experiencing Death (Kaplan-Meier Analysis)
Description: as for outcome 1
Time Frame: 6 months
Population: At the 6-month time point, 17 subjects had been censored and 4 had died, leaving 57 subjects "at risk" in the Kaplan-Meier freedom from mortality analysis at 6 months.
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 57
percentage of participants | 6.1

4. Primary Outcome: Percentage of Participants Experiencing Death (Kaplan-Meier Analysis)
Description: as for outcome 1
Time Frame: 12 months
Population: A total of 32 patients were analyzed because 41 subjects had been censored and 5 had died at 12 months time frame.
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 32
percentage of participants | 8.3

5. Secondary Outcome: Number of Participants With 0, 1, 2, and 3 MitraClip Devices Implanted
Description: This is one of the Device and Procedure-Related Endpoints. Implant Rate is defined as the rate of successful delivery and deployment of MitraClip device implant(s) with echocardiographic evidence of leaflet approximation and retrieval of the delivery catheter.
Time Frame: Day 0 (On the day of procedure)
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 78
Participants
  0 Mitra Clip devices | 1
  1 Mitra Clip devices | 41
  2 Mitra Clip devices | 35
  3 Mitra Clip devices | 1

6. Secondary Outcome: Number of Participants With Acute Procedural Success Rate
Description: Defined as successful MitraClip implantation with resulting MR of 2+ or less.
Time Frame: At day 0 (on the day of index procedure)
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 78
Participants | 39

7. Secondary Outcome: Procedure Time
Description: This is one of the Device and Procedure-Related Endpoints. Procedure Time is defined as the time elapsed from the start of the transseptal procedure to the time the Steerable Guide Catheter is removed.
Time Frame: At day 0 (on the day of index procedure)
Population: Procedure time was not available for 1 patient.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 77
Minutes | 133.5 (64.6)

8. Secondary Outcome: Device Time
Description: This is one of the Device and Procedure-Related Endpoints. Device Time is defined as the time the Steerable Guide Catheter is placed in the intra-atrial septum until the time the MitraClip Delivery System (CDS) is retracted into the Steerable Guide Catheter. Device Time is shorter in duration than Procedure Time because it does not include the time required to perform transseptal access into the left atrium.
Time Frame: At day 0 (on the day of index procedure)
Population: Device time was not available for 1 patient.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 77
Minutes | 91.2 (59.4)

9. Secondary Outcome: Fluoroscopy Duration
Description: This is one of the Device and Procedure-Related Endpoints. Mean fluoroscopy duration during the MitraClip procedure.
Time Frame: At day 0 (on the day of index procedure)
Population: Fluoroscopy duration was not available for 3 patient.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 75
Minutes | 41.2 (30.0)

10. Secondary Outcome: Total Contrast Volume
Description: This is one of the Device and Procedure-Related Endpoints.
Time Frame: At day 0 (on the day of index procedure)
Population: Total volume of contrast was not available for 5 patients.
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 73
Milliliters | 10.6 (29.3)

11. Secondary Outcome: Left Ventricle End Diastolic Volume (LVEDV)
Description: Left Ventricular end-diastolic volume (LVEDV) as determined by the core echo laboratory. Left Ventricular end-diastolic volume (LVEDV) measured using 2-dimensional echocardiography. The endocardium is traced at end-diastole (frame before mitral valve closure or maximum cavity dimension) in the 2- and 4-chamber views to calculate volumes.
Time Frame: At Baseline and Discharge (≤7 days of index procedure)
Population: A total of 65 patients had paired left ventricular end diastolic volume (LVEDV) measurements at both baseline and discharge. Thirteen patients had missing LVEDV at either baseline, discharge, or both time points.
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 65
Milliliters
  Baseline | 158.2 (68.4)
  Discharge | 151.3 (71.3)

12. Secondary Outcome: Left Ventricle End Diastolic Volume (LVEDV)
Description: as for outcome 11
Time Frame: At Baseline and 30 Days
Population: A total of 61 patients had paired left ventricular end diastolic volume (LVEDV) measurements at both baseline and 30 days. Six patients missed the 30-day visit and 11 patients had missing LVEDV at either baseline, the 30-day visit, or both time points.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 61
ml
  Baseline | 152.9 (67.8)
  30 Days | 148.2 (72.3)

13. Secondary Outcome: Left Ventricle End Diastolic Volume (LVEDV)
Description: as for outcome 11
Time Frame: At Baseline and 12 months
Population: A total of 41 patients were excluded from total analysis population as 5 patients died, 1 patient missed the 12-month visit, 6 patients had missing LVEDV at either baseline, the 12-month visit, or both time points, and finally 29 subjects 12-month visits were either expected or not due at the time that the ANZ trial was terminated.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 37
ml
  Baseline | 161.1 (75.7)
  12 Months | 150.1 (79.9)

14. Secondary Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: Left Ventricular end-systolic volume (LVESV) as determined by the core echo laboratory. Left Ventricular end-systolic volume (LVESV) measured using 2-dimensional echocardiography. The endocardium is traced at end-systole (frame prior to mitral valve opening or the minimum cavity area) in the 2- and 4-chamber views to calculate volumes.
Time Frame: At Baseline and Discharge (≤7 days of index procedure)
Population: A total of 65 patients had paired left ventricular end systolic volume (LVESV) measurements at both baseline and discharge. Thirteen patients had missing LVESV at either baseline, discharge, or both time points.
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 65
Milliliter
  Baseline | 93.3 (62.8)
  Discharge | 93.2 (63.3)

15. Secondary Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: as for outcome 14
Time Frame: At Baseline and 30 Days
Population: A total of 61 patients had paired left ventricular end systolic volume (LVESV) measurements at both baseline and 30 days. Six patients missed the 30-day visit and 11 patients had missing LVESV at either baseline, the 30-day visit, or both time points.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 61
ml
  Baseline | 88.5 (61.2)
  30 Days | 89.0 (61.7)

16. Secondary Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: as for outcome 14
Time Frame: At Baseline and 12 months
Population: Of total 78 subjects, 37 patients were analyzed because 5 patients died prior to the 12-month visit, 1 patient missed the 12-month visit, 6 patients had missing LVESV at either baseline, the 12-month visit, or both time points, and finally 29 patients 12-month visits were either expected or not due at the time that the ANZ trial was terminated.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 37
ml
  Baseline | 97.8 (70.4)
  12 Months | 91.7 (73.1)

17. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Left ventricular ejection fraction is assessed by transthoracic echocardiography according to Simpson's rule (biplane method of disks).
Time Frame: At Baseline and Discharge (≤7 days of index procedure)
Population: A total of 73 patients had paired left ventricular ejection fraction (LVEF) measurements at both baseline and discharge. Five patients had missing LVEF at either baseline, discharge, or both time points.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 73
percent
  Baseline | 47.2 (16.7)
  Discharge | 44.6 (16.3)

18. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: as for outcome 17
Time Frame: At Baseline and 30 Days
Population: A total of 67 patients had paired left ventricular ejection fraction (LVEF) measurements at both baseline and 30 days. Six patients missed the 30-day visit and 5 patients had missing LVEF at either baseline, the 30-day visit, or both time points.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 67
percent
  Baseline | 48.4 (16.3)
  30 Days | 46.5 (16.0)

19. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: as for outcome 17
Time Frame: At Baseline and 12 months
Population: A total of 40 patients included in analysis population because 5 patients died prior to the 12-month visit, 1 patient missed the 12-month visit, 3 patients had missing LVEF at either baseline, the 12-month visit, or both time points and 29 patients 12-month visits were either expected/not due at the time that the ANZ trial was terminated.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 40
percent
  Baseline | 46.9 (16.9)
  12 Months | 47.4 (18.8)

20. Secondary Outcome: Number of Participants With MR Severity
Description: Mitral regurgitation severity was determined based on the American Society of Echocardiography (ASE) Recommendations for Evaluation of The Severity of Native Valvular Regurgitation with Two-Dimensional and Doppler Echocardiography. MR severity was scored using the integrative method based on qualitative and quantitative echocardiographic parameters as described in the ASE guidelines.Site-assessed mitral regurgitation severity using echocardiography.
  MR severity was graded as follows: 0: None, 1+: Mild, 2+: Moderate, 3+: Moderate-to-Severe, 4+: Severe.
Time Frame: Baseline
Population: Mitral regurgitation severity is missing in 1 patient at Baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 77
Participants
  0: None | 0
  1+:Mild | 0
  2+: Moderate | 0
  3+: Moderate-to-Severe | 22
  4+: Severe | 55
  Not Evaluable | 0

21. Secondary Outcome: Number of Participants With MR Severity
Description: as for outcome 20
Time Frame: At discharge (≤7 days of index procedure)
Population: Mitral regurgitation severity is missing in 4 patient at Discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 74
Participants
  0: None | 1
  1+:Mild | 38
  2+: Moderate | 22
  3+: Moderate-to-Severe | 9
  4+: Severe | 3
  Not Evaluable | 1

22. Secondary Outcome: Number of Participants With MR Severity
Description: as for outcome 20
Time Frame: 30 days
Population: Mitral regurgitation severity is available for 69 patients at 30 days. Six patients missed the 30-day visit and 3 patients had not evaluated for MR severity at 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 69
Participants
  0: None | 1
  1+:Mild | 26
  2+: Moderate | 25
  3+: Moderate-to-Severe | 12
  4+: Severe | 5
  Not Evaluable | 0

23. Secondary Outcome: Number of Participants With MR Severity
Description: as for outcome 20
Time Frame: 6 months
Population: Mitral regurgitation severity is available for 60 patients at 6 months. Four patients died prior the 6-month visit, 1 patient missed the 6-month visit, 1 patient had missing MR severity at 6 months, and finally 12 patients 6-month visits were either expected or not due at the time that the ANZ trial was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 60
Participants
  0: None | 0
  1+:Mild | 20
  2+: Moderate | 24
  3+: Moderate-to-Severe | 12
  4+: Severe | 4
  Not Evaluable | 0

24. Secondary Outcome: Number of Participants With MR Severity
Description: as for outcome 20
Time Frame: 12 months
Population: Mitral regurgitation severity is available for 42 patients at 12 months. Five patients died prior the 12-month visit, 1 patient missed the 12-month visit, 1 patient had missing MR severity at 12 months, and finally 29 patients 12-month visits were either expected or not due at the time that the ANZ trial was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 42
Participants
  0: None | 2
  1+:Mild | 15
  2+: Moderate | 15
  3+: Moderate-to-Severe | 7
  4+: Severe | 3
  Not Evaluable | 0

25. Secondary Outcome: Left Ventricular Internal Diameter End Diastole (LVIDd)
Description: LVIDd is the measurements of the left ventricular internal dimension at end-diastole and normally corresponds to the largest cardiac dimension. LVIDd is measured by transthoracic echocardiography and the results are interpreted by the study's echocardiography core laboratory.
Time Frame: At Baseline and Discharge (≤7 days of index procedure)
Population: A total of 72 patients had paired left ventricular internal diameter in diastole (LVIDd) measurements at both baseline and discharge. Six patients had missing LVIDd at either baseline, discharge, or both time points.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 72
cm
  Baseline | 5.9 (1.0)
  Discharge | 5.7 (1.1)

26. Secondary Outcome: Left Ventricular Internal Diameter End Diastole (LVIDd)
Description: as for outcome 25
Time Frame: At Baseline and 30 Days
Population: A total of 67 patients had paired left ventricular internal diameter in diastole (LVIDd) measurements at both baseline and 30 days. Six patients missed the 30-day visit and 5 patients had missing LVIDd at either baseline, the 30-day visit, or both time points.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 67
cm
  Baseline | 5.9 (1.0)
  30 Days | 5.7 (1.0)

27. Secondary Outcome: Left Ventricular Internal Diameter End Diastole (LVIDd)
Description: as for outcome 25
Time Frame: At Baseline and 12 Months
Population: A total of 40 patients were included in analysis because 5 patients died prior to the 12-month visit,1 patient missed the 12-month visit,3 patients had missing LVIDd at either baseline,the 12-month visit,or both time points & 29 patients 12-month visits were either expected or not due at the time that the ANZ trial was terminated.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 40
cm
  Baseline | 6.0 (1.0)
  12 Months | 5.7 (1.1)

28. Secondary Outcome: Left Ventricular Internal Diameter End Systole (LVIDs)
Description: LVIDs is the measurements of the left ventricular internal dimension at end-systole and normally corresponds to the smallest cardiac dimension. LVIDs is measured by transthoracic echocardiography and the results are interpreted by the study's echocardiography core laboratory.
Time Frame: At Baseline and Discharge (≤7 days of index procedure)
Population: A total of 71 patients had paired left ventricular internal diameter in systole (LVIDs) measurements at both baseline and discharge. Seven patients had missing LVIDs at either baseline, discharge, or both time points.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 71
cm
  Baseline | 4.5 (1.4)
  Discharge | 4.4 (1.4)

29. Secondary Outcome: Left Ventricular Internal Diameter End Systole (LVIDs)
Description: as for outcome 28
Time Frame: At Baseline and 30 Days
Population: A total of 61 patients had paired left ventricular internal diameter in systole (LVIDs) measurements at both baseline and 30 days. Six patients missed the 30-day visit and 11 patients had missing LVIDs at either baseline, the 30-day visit, or both time points.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 61
cm
  Baseline | 4.5 (1.3)
  30 Days | 4.5 (1.3)

30. Secondary Outcome: Left Ventricular Internal Diameter End Systole (LVIDs)
Description: as for outcome 28
Time Frame: At Baseline and 12 Months
Population: A total of 36 patients had paired LVIDs measurements Because 5 patients died prior to the 12-month visit, 1 patient missed the 12-month visit, 7 patients had missing LVIDs at either baseline, the 12-month visit, or both time points and 29 patients 12-month visits were either expected or not due at the time that the ANZ trial was terminated.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 36
cm
  Baseline | 4.6 (1.4)
  12 Months | 4.5 (1.5)

31. Secondary Outcome: Regurgitant Volume
Description: Regurgitant volume as determined by the core echo laboratory. In the presence of regurgitation of one valve, without any intracardiac shunt, the flow through the affected valve is larger than through other competent valves. The difference between the two represents the regurgitant volume.
Time Frame: At Baseline and Discharge (≤7 days of index procedure)
Population: A total of 45 patients had paired regurgitant volume measurements at both baseline and discharge. Regurgitant volume data at either baseline, discharge, or both time points is missing for 33 patients.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 45
ml
  Baseline | 55.5 (31.2)
  Discharge | 25.1 (21.4)

32. Secondary Outcome: Regurgitant Volume
Description: as for outcome 31
Time Frame: At Baseline and 30 Days
Population: A total of 36 patients had paired regurgitant volume measurements at both baseline and 30 days. Six patients missed the 30-day visit and regurgitant volume data at either baseline, 30 days, or both time points is missing for 36 patients.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 36
ml
  Baseline | 61.9 (42.8)
  30 Days | 25.6 (28.5)

33. Secondary Outcome: Regurgitant Volume
Description: as for outcome 31
Time Frame: At Baseline and 12 Months
Population: A total of 20 patients were included in analysis because 5 patients died prior to the 12-month visit, 1 patient missed the 12-month visit, 23 patients have missing regurgitant volume data at either baseline, 12 months, or both time points & 29 patients 12-month visits were either expected or not due at the time that the ANZ trial was terminated.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 20
ml
  Baseline | 49.8 (29.0)
  12 Months | 73.3 (111.2)

34. Secondary Outcome: Regurgitant Fraction
Description: Regurgitant fraction as determined by the core echo laboratory. Regurgitant fraction is defined as the regurgitant volume divided by the forward stroke volume through the regurgitant valve.
Time Frame: At Baseline and Discharge (≤7 days of index procedure)
Population: A total of 18 patients had paired regurgitant fraction measurements at both baseline and discharge. Regurgitant fraction data at either baseline, discharge, or both time points is missing for 60 patients.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 18
Percentage
  Baseline | 38.9 (19.3)
  Discharge | 25.8 (36.5)

35. Secondary Outcome: Regurgitant Fraction
Description: as for outcome 34
Time Frame: At Baseline and 30 Days
Population: A total of 16 patients had paired regurgitant fraction measurements at both baseline and 30 days. Six patients missed the 30-day visit. Whereas, regurgitant fraction data at either baseline, 30 days, or both time points is missing for 56 patients.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 16
Percentage
  Baseline | 40.5 (19.7)
  30 Days | 15.2 (41.8)

36. Secondary Outcome: Regurgitant Fraction
Description: as for outcome 34
Time Frame: At Baseline and 12 Months
Population: Few patients excluded from analysis population because 5 patients died prior to the 12-month visit,1 patient missed the 12-month visit, 38 patients have missing regurgitant fraction data at either baseline, 12 months, or both time points and 29 patients 12-month visits were either expected or not due at the time that the ANZ trial was terminated.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 5
Percentage
  Baseline | 44.6 (15.9)
  12 Months | 36.8 (18.0)

37. Secondary Outcome: Mitral Valve Area (MVA) by Pressure Half-time (PHT)
Description: Measure of the area of the mitral valve orifice using transthoracic echocardiography. The pressure half time method is used to assess the presence and severity of mitral stenosis. Results are interpreted by the study's echocardiography core laboratory.
Time Frame: At Baseline and Discharge (≤7 days of index procedure)
Population: A total of 54 patients had paired mitral valve area (MVA) by pressure half-time measurements at both baseline and discharge. MVA data at either baseline, discharge, or both time points is missing for 24 patients.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 54
cm^2
  Baseline | 3.5 (1.2)
  Discharge | 2.4 (0.7)

38. Secondary Outcome: Mitral Valve Area (MVA) by Pressure Half-time (PHT)
Description: as for outcome 37
Time Frame: At Baseline and 30 Days
Population: A total of 50 patients had paired mitral valve area (MVA) by pressure half-time measurements at both baseline and 30 days. Six patients missed the 30-day visit. Where as, regurgitant fraction data at either baseline, 30 days, or both time points is missing for 22 patients.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 50
cm^2
  Baseline | 3.5 (1.0)
  30 Days | 2.3 (0.7)

39. Secondary Outcome: Mitral Valve Area (MVA) by Pressure Half-time (PHT)
Description: as for outcome 37
Time Frame: At Baseline and 12 Months
Population: A total of 29 patients were analyzed because 5 patients died prior to the 12-month visit,1 patient missed the 12-month visit, 14 patients have missing MVA data at either baseline, 12 months, or both time points. Finally 29 patients 12-month visits were either expected or not due at the time that the ANZ trial was terminated.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 29
cm^2
  Baseline | 3.8 (1.4)
  12 Months | 2.3 (0.7)

40. Secondary Outcome: Mitral Valve Mean Gradient
Description: Mitral valve mean gradient is defined as the mean pressure gradients across the mitral valve as measured by echocardiography.
Time Frame: At Baseline and Discharge (≤7 days of index procedure)
Population: A total of 65 patients had paired mitral valve mean gradient (MVG) measurements at both baseline and discharge. MVG data at either baseline, discharge, or both time points is missing for 13 patients.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 65
mmHg
  Baseline | 2.3 (1.0)
  Discharge | 3.7 (1.6)

41. Secondary Outcome: Mitral Valve Mean Gradient
Description: as for outcome 40
Time Frame: At Baseline and 30 Days
Population: A total of 59 patients had paired mitral valve mean gradient (MVG) measurements at both baseline and 30 days. Six patients missed the 30-day visit. MVG data at either baseline, 30 days, or both time points are missing for 13 patients.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 59
mmHg
  Baseline | 2.3 (1.0)
  30 Days | 3.5 (1.7)

42. Secondary Outcome: Mitral Valve Mean Gradient
Description: as for outcome 40
Time Frame: At Baseline and 12 Months
Population: A total of 34 patients had paired MVG measurements because 5 patients died prior to the 12-month visit, 1 patient missed the 12-month visit, 9 patients have missing MVG data at either baseline, 12 months, or both time points. Finally 29 patients 12-month visits were either expected or not due at the time that the ANZ trial was terminated.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 34
mmHg
  Baseline | 2.3 (1.0)
  12 Months | 3.4 (1.4)

43. Secondary Outcome: Left Atrial Volume
Description: Left atrial volume is assessed by echocardiography. Using the single plane method of disks, the left atrial volume is derived by planimetry in the 4-chamber view at end-systole.
Time Frame: At Baseline and Discharge (≤7 days of index procedure)
Population: A total of 67 patients had paired left atrial (LA) volume measurements at both baseline and discharge. LA volume data at either baseline, discharge, or both time points are missing for 11 patients.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 67
ml
  Baseline | 141.7 (54.7)
  Discharge | 141.8 (62.9)

44. Secondary Outcome: Left Atrial Volume
Description: as for outcome 43
Time Frame: At Baseline and 30 Days
Population: A total of 62 patients had paired left atrial (LA) volume measurements at both baseline and 30 days. Six patients missed the 30-day visit, Where as LA volume data at either baseline, 30 days, or both time points are missing for 10 patients.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 62
ml
  Baseline | 140.4 (54.3)
  30 Days | 138.8 (58.6)

45. Secondary Outcome: Left Atrial Volume
Description: as for outcome 43
Time Frame: At Baseline and 12 Months
Population: A total of 39 patients had paired LA volume measurements because 5 patients died prior to the 12-month visit, 1 patient missed the 12-month visit, 4 patients have missing LA volume data at either baseline, 12 months, or both time points and 29 patients 12-month visits were either expected or not due at the time that the ANZ trial was terminated.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 39
ml
  Baseline | 148.5 (59.0)
  12 Months | 132.4 (64.5)

46. Secondary Outcome: Six Minute Walking Distance
Description: The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. It is a measure of a patient's exercise capacity.
Time Frame: Baseline
Population: Six-minuted walk test (6MWT) distance is available for 76 patients at baseline because 2 patients did not complete the 6MWT at baseline.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 76
Meters | 271.0 (119.4)

47. Secondary Outcome: Six Minute Walking Distance
Description: as for outcome 46
Time Frame: 30 days
Population: Six-minuted walk test (6MWT) distance is available for 68 patients at 30 days. Six patients missed the 30-day visit and 4 patients did not complete the 6MWT at 30-days.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 68
Meters | 297.3 (130.7)

48. Secondary Outcome: Six Minute Walking Distance
Description: as for outcome 46
Time Frame: 6 months
Population: Six-minuted walk test (6MWT) distance is available for 60 patients at 6 months. Four patients died prior to the 6-month visit, 1 patient missed the 6-month visit, 1 patient did not complete the 6MWT at 6-months, and finally, 12 patients 6-month visits were either expected or not due at the time that the ANZ trial was terminated.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 60
Meters | 324.3 (139.5)

49. Secondary Outcome: Six Minute Walking Distance
Description: as for outcome 46
Time Frame: 12 months
Population: Six-minuted walk test (6MWT) distance is available for 39 patients at 12 months. Five patients died prior to the 12-month visit, 1 patient missed the 12-month visit, 4 patients did not complete the 6MWT at 12 months, and finally 29 patients 6-month visits were either expected or not due at the time that the ANZ trial was terminated.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 39
Meters | 329.9 (120.8)

50. Secondary Outcome: Percentage of Participants With New York Heart Association (NYHA) Class
Description: * Class I Patients with cardiac disease but without resulting limitations of physical activity;
  * Class II Patients with cardiac disease resulting in slight limitation of physical activity. Patients are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain;
  * Class III Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary physical activity causes fatigue, palpitation dyspnea, or anginal pain;
  * Class IV Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 78
percentage of participants
  NYHA I | 2.6
  NYHA II | 26.9
  NYHA III | 51.3
  NYHA IV | 19.2

51. Secondary Outcome: Percentage of Participants With New York Heart Association (NYHA) Class
Description: as for outcome 50
Time Frame: 30 days
Population: A total of 69 patients were included in analysis population because 6 patients had lost-to-follow up at 30 days and 3 patients did not have a NYHA functional class assessment.
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 69
percentage of participants
  NYHA I | 36.2
  NYHA II | 44.9
  NYHA III | 15.9
  NYHA IV | 2.9

52. Secondary Outcome: Percentage of Participants With New York Heart Association (NYHA) Class
Description: as for outcome 50
Time Frame: 6 months
Population: NYHA functional class assessment is available for 60 patients at 6 months. Four patients died prior to the 6-month visit, 1 patient missed the 6-month visit, 1 patient did not have a NYHA functional class assessment at 6-months, and finally 12 patients 6-month visits were either expected or not due at the time that the ANZ trial was terminated.
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 60
percentage of participants
  NYHA I | 33.3
  NYHA II | 56.7
  NYHA III | 8.3
  NYHA IV | 1.7

53. Secondary Outcome: Percentage of Participants With New York Heart Association (NYHA) Class
Description: as for outcome 50
Time Frame: 12 months
Population: NYHA functional class assessment is available for 40 patients at 12 months.Five patients died prior to the 12-month visit,1 patient missed the 12-month visit, 3 patients did not have a NYHA functional class assessment and finally 29 patients 12-month visits were either expected or not due at the time that the ANZ trial was terminated.
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 40
percentage of participants
  NYHA I | 52.5
  NYHA II | 42.5
  NYHA III | 2.5
  NYHA IV | 2.5

54. Secondary Outcome: Change in Minnesota Living With Heart Failure (MLWHF) Quality of Life (QOL) Score From Baseline to 30 Days
Description: The Minnesota Living with Heart Failure Questionnaire(MLHFQ) is comprised of 21 questions.The response for each question ranges from 0(no affect on the patient's living) to 5(affected the patient's life very much during the past month).The total score for the 21 items can range from 0-105.A lower&higher MLHFQ score indicates less effect of heart failure&the worse impact of heart failure on a patient's QOL,respectively.Although the MLHFQ incorporates relevant aspects of the key dimensions of QOL (physical and emotional),the questionnaire was not designed to measure any particular dimension separately.The total score should be taken as the best measure of how heart failure and treatments impact QOL.
  The total score is the sum of a)the physical dimension,measured using 8 questions (possible subscale score range 0-40) b)the emotional dimension,measured using 5 questions(possible subscale score from 0-25)&c) other factors,measured using 8 questions (possible subscale score from 0-40).
Time Frame: 30 days
Population: Paired Minnesota Living with Heart Failure Questionnaire (MLHFQ) quality of life data was available for 70 patients at Baseline and 30 days. Six patients missed their 30-day visit and 2 patients did not complete the MLHFQ at either baseline, 30 days, or both time points.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 70
scores on a scale
  Baseline | 50.4 (23.2)
  30 days | 26.4 (20.1)
  Difference (30 days - Baseline) | -24.0 (21.6)

55. Secondary Outcome: Change in Minnesota Living With Heart Failure (MLWHF) Quality of Life (QOL) Score From Baseline to 6 Months
Description: as for outcome 54
Time Frame: 6 months
Population: Paired Minnesota Living with Heart Failure Questionnaire (MLHFQ) quality of life data was available for 61 patients at Baseline and 6 months. Four patients died prior to the 6-month visit,1 patient missed the 6-month visit and 12 patients 6-month visits were either expected or not due at the time that the ANZ trial was terminated.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 61
scores on a scale
  Baseline | 49.5 (23.5)
  6 months | 28.0 (21.3)
  Difference (6 months - Baseline) | -21.5 (22.5)

56. Secondary Outcome: Change in Minnesota Living With Heart Failure (MLWHF) Quality of Life (QOL) Score From Baseline to 12 Months
Description: as for outcome 54
Time Frame: 12 months
Population: Paired MLHFQ quality of life data was available for 40 patients at Baseline and 12 months.Five patients died prior to the 12-month visit,1 patient missed the 12-month visit,3 patients did not complete the MLHFQ assessment. Finally, 29 patients 12-month visits were either expected or not due at the time that the ANZ trial was terminated.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 40
scores on a scale
  Baseline | 51.1 (25.1)
  12 months | 30.2 (22.7)
  Difference (12 months - Baseline) | -20.9 (25.5)

57. Secondary Outcome: Percentage of Participants Experiencing Freedom From Death and Congestive Heart Failure (Kaplan-Meier Curve Analysis)
Description: Death: Defined as all causes of death for the primary safety Major Adverse Event (MAE) Endpoint.
  Death is further divided into 2 categories:
  A. Cardiac death is defined as death due to any of the following:
  * Acute myocardial infarction
  * Cardiac perforation/pericardial tamponade
  * Arrhythmia or conduction abnormality
  * Stroke within 30 days of the procedure or stroke suspected of being related to the procedure
  * Death due to any complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery
  * Any death for which a cardiac cause cannot be excluded.
  B. Non-cardiac death is defined as a death not due to cardiac causes (as defined above).
  Congestive Heart Failure (CHF): Defined as a documented diagnosis of CHF on the hospital admission report or discharge summary.
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 78
percentage of participants | 100

58. Secondary Outcome: Percentage of Participants Experiencing Freedom From Death and Congestive Heart Failure (Kaplan-Meier Curve Analysis)
Description: as for outcome 57
Time Frame: 30 days
Population: Two patient were lost to follow-up at the 30-day time point and 1 had been censored at Baseline. Therefore, 73 patients were included in the "at risk" population in the Kaplan-Meier freedom from death and congestive heart failure analysis at 30 days.
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 73
percentage of participants | 96.1

59. Secondary Outcome: Percentage of Participants Experiencing Freedom From Death and Congestive Heart Failure (Kaplan-Meier Curve Analysis)
Description: as for outcome 57
Time Frame: 6 months
Population: At 6 months, 55 patients were considered "at risk" because 17 had been censored, and 6 patients experienced an event (i.e. death or CHF event).
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 55
percentage of participants | 91.5

60. Secondary Outcome: Percentage of Participants Experiencing Freedom From Death and Congestive Heart Failure (Kaplan-Meier Curve Analysis)
Description: as for outcome 57
Time Frame: 12 months
Population: At 12 months, 31 patients were considered "at risk" because 38 had been censored and 9 patients experienced an event (i.e. death or CHF event).
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 31
percentage of participants | 85.3

61. Secondary Outcome: Number of Participants With Mitral Valve Surgery
Description: Mital Valve Surgery Post-MitraClip Procedure; Surgery Types includes Replacement and Repair.
Time Frame: 30 days of Post-MitraClip Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 78
Participants
  Recurring mitral regurgitation | 1
  Device failure | 1

62. Secondary Outcome: Number of Participants With Second Intervention to Place an Additional MitraClip Device
Description: Second MitraClip device interventions are reported by Abbott Vascular personnel on Procedural Observation Forms. A second MitraClip device intervention is a good option for patients with MR following placement of the original MitraClip device.
Time Frame: Through 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 78
Participants
  Recurring mitral regurgitation | 2
  Single leaflet device attachment (SLDA) | 1

63. Secondary Outcome: Rate of Patients Rehospitalized
Description: Defined as re-admission of patients to the hospital following discharge from the Clip procedure.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 78
Participants
  All re-hospitalizations | 35
  Heart Failure-related re-hospitalizations | 10
  Other cardiac-related re-hospitalizations | 11
  Other non-cardiac-related re-hospitalizations | 22

64. Secondary Outcome: Duration of Rehospitalization
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 78
Days
  All re-hospitalizations | 8.4 (12.9)
  Heart Failure-related re-hospitalizations | 18.38 (20.65)
  Other cardiac-related re-hospitalizations | 2.87 (5.03)
  Other non-cardiac-related re-hospitalizations | 7.44 (9.01)

65. Secondary Outcome: Number of Participants at Discharge Facility
Description: This is the economic data reported to support the MitraClip System economic analysis.
Time Frame: < or = 12 days
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 78
Participants
  Home | 70
  Home with home health care | 4
  Skilled nursing facility | 1
  Nursing home | 0
  Death | 2
  Other | 1

66. Secondary Outcome: Post-procedure Intensive Care Unit (ICU)/Critical Care Unit (CCU)/Post-anesthesia Care Unit (PACU) Duration
Description: ICU and hospital stay is defined as the mean duration of time that patients spent in the ICU (Intensive Care Unit)/ CCU (Cardiac Care Unit)/ PACU (Post-Anesthesia Care Unit) following the MitraClip procedure.
Time Frame: Post index procedure within 30 days
Population: Post-Procedure ICU/CCU/PACU duration was not available for 4 patients.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 74
Hours | 62.1 (85.7)

67. Secondary Outcome: Post-procedure Hospital Stay
Description: This is the Economic data reported to support the MitraClip System economic analysis. It is defined as the mean duration of time that patients spent in hospital following the MitraClip procedure.
Time Frame: Post index procedure within 30 days
Population: Duration of post-procedure hospital stay was not available for 3 patients.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MitraClip Implant
Number analyzed (Participants) | 75
Days | 3.4 (2.2)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | MitraClip Implant
All-Cause Mortality (participants affected / at risk) | 0/78
Serious Adverse Events (participants affected / at risk) | 37/78
Other Adverse Events (participants affected / at risk) | 52/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MitraClip Implant (N=78)
Angina/Chest Pain (Cardiac disorders) | 2 (2)
Arrhythmias (Cardiac disorders) | 6 (12)
Bleeding (Vascular disorders) | 5 (6)
Fever or Hyperthermia (General disorders) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 2 (2)
Hypotension/Hypertension (Vascular disorders) | 4 (4)
Mitral Valve/Leaflet Injury (Injury, poisoning and procedural complications) | 2 (2)
Other (General disorders) | 25 (38)
Renal Insufficiency or Failure (Renal and urinary disorders) | 5 (5)
Respiratory Failure/Atelectasis/Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Septicemia (Infections and infestations) | 2 (3)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Stroke (Cardiac disorders) | 3 (3)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MitraClip Implant (N=78)
Angina/Chest Pain (Cardiac disorders) | 5 (7)
Arrhythmias (Cardiac disorders) | 10 (19)
Bleeding (Vascular disorders) | 24 (35)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Fever or Hyperthermia (General disorders) | 3 (3)
Hematoma (Vascular disorders) | 19 (28)
Hypotension/Hypertension (Vascular disorders) | 8 (9)
Infection at Access Site (Infections and infestations) | 1 (1)
Mitral Valve/Leaflet Injury (Infections and infestations) | 3 (3)
Nausea/Vomiting (General disorders) | 6 (7)
Other (General disorders) | 47 (136)
Pain at Incision Site (General disorders) | 4 (4)
Renal Insufficiency or Failure (Renal and urinary disorders) | 5 (5)
Respiratory Failure/Atelectasis/Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Septicemia (Infections and infestations) | 2 (3)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Stroke (Cardiac disorders) | 3 (3)
Urinary Tract Infection (Renal and urinary disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less